CLINICAL TRIAL: NCT03820479
Title: An Observational Study to Investigate Quality of Recovery, the Incidence and Impact of Post-Operative Nausea and Vomiting (PONV)/Post-Discharge Nausea and Vomiting (PDNV) up to Day 7 in Females Undergoing Laparoscopic Abdominal Surgery Provided Apfel-score Based PONV Care and Prophylaxis
Brief Title: A Study to Investigate Quality of Recovery up to Day 7 in Females Undergoing Laparoscopic Abdominal Surgery Provided Apfel-score Based PONV Care and Prophylaxis
Status: Completed | Type: Observational
Sponsor: Danderyd Hospital (Other)
Responsible Party: Principal Investigator, EmmaObrink, Principal Investigator, Danderyd Hospital
Other Study IDs: DanderydH
Record Dates: First submitted 2019-01-23; First posted 2019-01-29 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2024-10

CONDITIONS: Quality of Recovery
Keywords: Quality of recovery; PONV; PDNV
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Clinical Protocols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Apfel score 1: Female
  Interventions: Other: Protocol
- Apfel score 2: Female, non smoker
  Interventions: Other: Protocol
- Apfel score 3: Female, non smoker, under 40 years old
  Interventions: Other: Protocol
- Apfel score 4: Female, non smoker, under 40 years old, previous history of PONV
  Interventions: Other: Protocol

INTERVENTIONS:
Other: Protocol — Best practice of protocol

SUMMARY:
SYNOPSIS Title: An observational study to investigate Quality of Recovery and the incidence and impact of Post-Operative Nausea and Vomiting (PONV)/Post-Discharge Nausea and Vomiting (PDNV) and up to 7 days in females undergoing laparoscopic abdominal surgery provided Apfel-score based PONV care and prophylaxis.

Study period: September 2018- September 2019

Hypothesis: When a high risk patient, Apfel-score 3 or 4, is given Apfel-score based PONV care with strict adherence to PONV guidelines there should be no difference in Quality of Recovery between a high-risk patient and a low-risk patient.

Aim: The aim of the study is to investigate if it is possible to reach no difference in Quality of Recovery (QoR) between a high-risk patient and a low risk patient using Apfel-score based PONV care.

Primary objective: Assessing Quality of Recovery, using QoR15 at 24h, 48h, 72h and after 7 days.

Secondary objectives: Assessing the incidence and severity of PONV and PDNV in females undergoing laparoscopic surgery up to 72h. Assessing PONV and PDNV severity and duration. Nicotine habits and impact on PONV.

Study outline: Females scheduled for elective abdominal laparoscopic surgery will be provided PONV care based on Apfel risk-score. All patients will fill in the QoR15 form before surgery (base line). PONV and PDNV will be assessed in the PACU postoperatively, after 24h, 48h and 72h. Quality of Recovery will be assessed up to 7 days after surgery.

Treatment: The females will be given ordinary care after local routines, with strict adherence to PONV guidelines.

Study population: 100 females aged 18-65, ASA 1-2, undergoing laparoscopic abdominal surgery in Danderyds Hospital.

Primary outcome variables and examinations: When the QoR 15 reaches base line or better after surgery. Number of times the females experience nausea, retching or vomiting and the impact of emetic symptoms on the QoR.

ELIGIBILITY:
Inclusion Criteria:

* ASA class 1-2

Exclusion Criteria:

* ASA 4, obese

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Female undergoing laparoscopic surgery
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Quality of recovery, QoR15 (Quality of Recovery 15) | 7 days
  Score, a valid questionnaire to measure quality of recovery, 15 questions, maximum score 150p. VAS scales for each items; 0 bad score, 10 optimal score. Mean values for group, sum score will be compared with parametric tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Danderyds Sjukhus, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No